CLINICAL TRIAL: NCT05529004
Title: Preoperative Pregabalin to Prevent Postoperative Nausea & Vomiting in Laparoscopic Surgery.
Brief Title: A 6 Months Double Blind Trial to Prevent PONV in Laparoscopic Cholecystectomy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Al Safwa University College (Other)
Responsible Party: Principal Investigator, Mohammed AbdulZahra Sasaa, Anesthetist, Al Safwa University College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: pregabalin and PONV
Record Dates: First submitted 2022-08-30; First posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: nausea, vomiting, cholecystectomy, oral pregapalin
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting | interventions — Anesthesia, General; Laparoscopes

STUDY DESIGN:
Intervention Model Description: Randomized Double Blind study.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Preoperative pregabalin to prevent postoperative nausea & vomiting in laparoscopic surgery. (Experimental): participants receive pregapalin 75mg cap orally 30 min before surgery
  Interventions: Drug: Oral Capsule pregapalin; Device: laparoscope device
- placebo (No Intervention): participants hasn't receive pregapalin capsule

INTERVENTIONS:
Drug: Oral Capsule pregapalin — oral cap of pregapalin has been administration to patient before surgery to prvent PONV
  Other Names: general anesthesia
  Arms: Preoperative pregabalin to prevent postoperative nausea & vomiting in laparoscopic surgery.
Device: laparoscope device — general anesthesia with complete relaxation under laparoscopic cholecystectomy
  Arms: Preoperative pregabalin to prevent postoperative nausea & vomiting in laparoscopic surgery.

SUMMARY:
As long as anesthesia is administered, postoperative nausea and vomiting (PONV) will continue to be a frequent and upsetting comorbidity. Vomiting and nausea can significantly slow down recovery, raise staffing and drug expenses, and decrease patient satisfaction during perioperative procedures.

Nausea it is a conscious recognition of subconscious excitation in area of medulla closely associated with or a part of the vomiting center, or it is sensation of discomfort at upper abdomen and unease sensation with involuntary order to vomit. While vomiting It is a mean by which the upper GIT rides of its contents when any part of upper GIT becomes irritated, over distended or over excitable.

The PONV is the most feared postoperative symptoms & it may impaired dressing , surgical repairs & increased ( bleeding , pain , risk of gastric contents aspiration ) & if it is prolonged will leads to electrolytes , fluid imbalance & dehydration ; the PONV can occurs after up to 90 % of operative procedures ; The common risk factors of PONV are : young age , female gender, history of ( PONV , motion sickness ) , those not smokers , early mobilization after surgery , early drinking & eating after operations , procedures like (laparoscopic , gynecological , abdominal , ENT , squint ) , postoperative severe pain , narcotic premedication , possibly prolonged general anesthesia , gastric distention , stimulation of the pharynx , hypoxemia , hypotension , & dehydration.

The PONV can reduced by: avoidance of triggers where possible, uses of anti-emetics drugs, techniques & procedures associated with low incidence of PONV (e.g. propofol) & give intravenous fluids; with prophylaxis the incidence is usually under 30% in high risk cases, the most effective approach for prevention of PONV is the use of multiple strategies & different drugs.

The pregabalin (C8H17NO2), is a newer drug & recently introduced at 1990. as anticonvulsive medication. We evaluated the effect of oral pregabalin on postoperative nausea and vomiting in laparoscopic cholecystectomy cases.

DETAILED DESCRIPTION:
Pregabalin has been found to minimize the need for opioid as well as non-steroid anti-inflammatory medications and relieve pain with different type of surgery, along with consideration of a diverse mechanisms, preoperative oral pregabalin has been reported to have antiemetic effect postoperatively. postoperative laparoscopic cholecystectomy, are associated with nausea and Vomiting and it's a concern that dictates the need for antiemetic which gives intravenously; as the intravenous drugs with intravenous fluid is becoming more common, the use of oral pregabalin is frequently mentioned, on the other hand, the intravenous antiemetic medication has some side effect.

Aim of the study:

To evaluate the effect of oral pregabalin on postoperative nausea and vomiting in laparoscopic cholecystectomy cases.

Design: Randomized Double Blind study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 - < 55 years.
* Both gender (male & female).
* Patients ASA physical status1.
* Procedures with high risk of postoperative nausea & vomiting.
* Elective operations under general anesthesia with laparoscopic cholecystectomy.

Exclusion Criteria:

* Age ≥ 55 years.
* Emergency operations,
* Patient refusal, allergy to pregabalin.
* Pregnant patients, patients taken preoperative anti-emetic medications.
* Patients with cardiac respiratory endocrine diseases.
* Total intravenous maintenance general anesthesia and thiopental as induction agent.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Preoperative Pregabalin to Prevent Postoperative Nausea & Vomiting in Laparoscopic Surgery. | Baseline
  Analysis of pregabalin group compare with the control group in laparoscopic cholecystectomy patients. to fined effective of oral pregapaline on PONV. we assess the incidence of postoperative nausea and vomiting by the use of Koivuranta Score.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Habib AS, Gan TJ. Evidence-based management of postoperative nausea and vomiting: a review. Can J Anaesth. 2004 Apr;51(4):326-41. doi: 10.1007/BF03018236. PMID 15064261
- [Background] Koivuranta MK, Laara E, Ryhanen PT. Antiemetic efficacy of prophylactic ondansetron in laparoscopic cholecystectomy. A randomised, double-blind, placebo-controlled trial. Anaesthesia. 1996 Jan;51(1):52-55. doi: 10.1111/j.1365-2044.1996.tb07654.x. PMID 8669567
- [Background] Gan TJ, Belani KG, Bergese S, Chung F, Diemunsch P, Habib AS, Jin Z, Kovac AL, Meyer TA, Urman RD, Apfel CC, Ayad S, Beagley L, Candiotti K, Englesakis M, Hedrick TL, Kranke P, Lee S, Lipman D, Minkowitz HS, Morton J, Philip BK. Fourth Consensus Guidelines for the Management of Postoperative Nausea and Vomiting. Anesth Analg. 2020 Aug;131(2):411-448. doi: 10.1213/ANE.0000000000004833. PMID 32467512
- [Result] Habib AS, Chen YT, Taguchi A, Hu XH, Gan TJ. Postoperative nausea and vomiting following inpatient surgeries in a teaching hospital: a retrospective database analysis. Curr Med Res Opin. 2006 Jun;22(6):1093-9. doi: 10.1185/030079906X104830. PMID 16846542
- [Result] Carroll NV, Miederhoff PA, Cox FM, Hirsch JD. Costs incurred by outpatient surgical centers in managing postoperative nausea and vomiting. J Clin Anesth. 1994 Sep-Oct;6(5):364-9. doi: 10.1016/s0952-8180(05)80004-2. PMID 7986507
- [Result] Metz A, Hebbard G. Nausea and vomiting in adults--a diagnostic approach. Aust Fam Physician. 2007 Sep;36(9):688-92. PMID 17885699